CLINICAL TRIAL: NCT03530306
Title: Treatment Evaluation of Neuromodulation for Tinnitus - Stage A2 (TENT-A2)
Brief Title: Treatment Evaluation of Neuromodulation for Tinnitus - Stage A2
Acronym: TENT-A2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromod Devices Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Neuromoddevices TENT-A2
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PS1-PS4 (Active Comparator)
  Interventions: Device: PS1-PS4
- PS6-PS10 (Active Comparator)
  Interventions: Device: PS6-PS10
- PS7-PS4 (Active Comparator)
  Interventions: Device: PS7-PS4
- PS9-PS6 (Active Comparator)
  Interventions: Device: PS9-PS6

INTERVENTIONS:
Device: PS1-PS4 — Participants in this arm shall be given PS1 during the first half of treatment and PS4 during the second half of treatment. During the expected 12-week treatment period, the participants will be presented with audio stimuli and electrical pulses for somatosensory stimulation.
  Arms: PS1-PS4
Device: PS6-PS10 — Participants in this arm shall be given PS6 during the first half of treatment and PS10 during the second half of treatment. During the expected 12-week treatment period, the participants will be presented with audio stimuli and electrical pulses for somatosensory stimulation.
  Arms: PS6-PS10
Device: PS7-PS4 — Participants in this arm shall be given PS7 during the first half of treatment and PS4 during the second half of treatment. During the expected 12-week treatment period, the participants will be presented with audio stimuli and electrical pulses for somatosensory stimulation.
  Arms: PS7-PS4
Device: PS9-PS6 — Participants in this arm shall be given PS9 during the first half of treatment and PS6 during the second half of treatment. During the expected 12-week treatment period, the participants will be presented with audio stimuli and electrical pulses for somatosensory stimulation.
  Arms: PS9-PS6

SUMMARY:
This is a four arm, patient subtyping and parameter optimisation study for a neuromodulation treatment for tinnitus.

DETAILED DESCRIPTION:
Participants with chronic tinnitus will be provided with a CE marked neuromodulation device. Participants are randomized to one of four different treatment arms. The treatment period is intended for 12 weeks of use. Based on the clinical investigation plan, participants are informed that their stimulation settings can change between the first and second halves of the treatment period and that the differences may be perceptually noticeable. Differences in tinnitus severity scores will be compared between and within treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Ability to read and understand English
* Willing and able to provide informed consent
* Willing to commit to the full duration of the study
* Baseline Tinnitus Handicap Inventory (THI) score of >= 38 points
* Subjective tinnitus of 3 months to 10 years
* Maximum AC pure-tone audiometry hearing loss of 80 dB HL in any test frequency in the set {2,3,4,6,8}kHz or 40 dB HL in the set {250,500,1000}Hz either unilaterally or bilaterally
* Baseline Minimum Masking Level (MML) of 20 to 80 dB HL
* Tonal tinnitus

Exclusion Criteria:

* Diagnosed with objective tinnitus
* Commenced usage of hearing aid within the last 90 days
* Cases where pulsatility is the dominant feature of tinnitus
* Patients whose tinnitus cannot be masked during Minimum Masking Level (MML) assessment
* Meniere's disease
* Significantly severe Loudness Discomfort Level (LDL, less than 30 dB SL)
* Depression or neuro-psychological condition, previously diagnosed or identified from the State-Trait Anxiety Inventory (STAI) with score greater than 120
* Diagnosed with somatic tinnitus resulting from head or neck injury
* Temporomandibular Joint Disorder (TMJ)
* Current or previous involvement in medico-legal cases
* Pregnancy
* Oral piercings
* Neurological condition that may lead to loss of consciousness (e.g. epilepsy) or is considered to be the dominant feature of the tinnitus, as assessed by audiologist or ENT consultant
* Severe cognitive impairment based on Mini Mental State Examination (MMSE, less than 20)
* Patient with a pacemaker or other electro-active implanted device
* Have used Neuromod Devices products in the past
* Participants currently prescribed drugs for a central nervous system pathology, i.e. epilepsy, Multiple Sclerosis (MS), Parkinson's, bi-polar disorder
* The site Principal Investigator does not deem the candidate to be suitable for the study for other reasons not listed above
* Self-reporting episodes of auditory hallucinations
* Abnormal Otoscopy as assessed by the Audiologist, including active Otitis Media, perforation and hearing loss that is identified as completely conductive
* Abnormal Tympanometry as assessed by the Audiologist

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | Between-arm and within-arm changes in THI after 6 weeks of treatment

OTHER OUTCOMES:
Tinnitus Handicap Inventory (THI) | Between-arm and within-arm changes in THI after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Brendan Conlon, Principal Investigator — St. James's Hospital, Ireland
Locations (1):
- St. James's Wellness Trust Clinical Research Facility, Dublin, Ireland

REFERENCES:
- [Background] Conlon B, Hamilton C, Hughes S, Meade E, Hall DA, Vanneste S, Langguth B, Lim HH. Noninvasive Bimodal Neuromodulation for the Treatment of Tinnitus: Protocol for a Second Large-Scale Double-Blind Randomized Clinical Trial to Optimize Stimulation Parameters. JMIR Res Protoc. 2019 Sep 27;8(9):e13176. doi: 10.2196/13176. PMID 31573942
- [Result] Conlon B, Hamilton C, Meade E, Leong SL, O Connor C, Langguth B, Vanneste S, Hall DA, Hughes S, Lim HH. Different bimodal neuromodulation settings reduce tinnitus symptoms in a large randomized trial. Sci Rep. 2022 Jun 30;12(1):10845. doi: 10.1038/s41598-022-13875-x. PMID 35773272